CLINICAL TRIAL: NCT00989781
Title: Mechanisms of Increased Androgen Production Among Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Jeffrey Chang, MD, Principal Investigator, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 090560
Record Dates: First submitted 2009-10-05; First posted 2009-10-06 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS, Androgens, ovary, polycystic
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Chorionic Gonadotropin; Ovidrel; follitropin alfa; Adrenocorticotropic Hormone; Cosyntropin; Dexamethasone; Adrenal Cortex Hormones; Glucose; Sugars

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCOS women (Experimental): Each subject will undergo pelvic 3D ultrasound followed by an iv recombinant human chorionic gonadotropin (r-hCG) stimulation test. One month later the r-hCG test will be repeated 24 hr after an injection of recombinant human follicle stimulating hormone (FSH).
  After 1 month, subjects will receive a 7 hr dose-response infusion of adrenocorticotropin (ACTH) with blood sampling. Dexamethasone will be given prior to ACTH.
  After 1 month, subject will receive r-hCG as described above followed the next day by an oral glucose tolerance test (OGTT). Subsequently, subjects will take Diazoxide 3 times a day for 2 weeks. At weekly intervals (2 weeks), the r-hCG stimulation test will be repeated followed the next day by an OGTT as described above.
  Interventions: Radiation: 3-D Ultrasound; Drug: recombinant human chorionic gonadotropin; Drug: Recombinant human follicle stimulating hormone; Drug: Adrenocorticotropin; Drug: Dexamethasone; Drug: Glucose
- Normal women (Experimental): Each subject will undergo pelvic 3D ultrasound followed by an iv recombinant human chorionic gonadotropin (r-hCG) stimulation test. One month later the r-hCG test will be repeated 24 hr after an injection of recombinant human follicle stimulating hormone (FSH).
  After 1 month, subjects will receive a 7 hr dose-response infusion of adrenocorticotropin (ACTH) with blood sampling. Dexamethasone will be given prior to ACTH.
  After 1 month, subject will receive r-hCG as described above followed the next day by an oral glucose tolerance test (OGTT). Subsequently, subjects will take Diazoxide 3 times a day for 2 weeks. At weekly intervals (2 weeks), the r-hCG stimulation test will be repeated followed the next day by an OGTT as described above.
  Interventions: Radiation: 3-D Ultrasound; Drug: recombinant human chorionic gonadotropin; Drug: Recombinant human follicle stimulating hormone; Drug: Adrenocorticotropin; Drug: Dexamethasone; Drug: Glucose

INTERVENTIONS:
Radiation: 3-D Ultrasound — One time pelvic ultrasound
Drug: recombinant human chorionic gonadotropin — Recombinant human chorionic gonadotropin will be given iv and blood samples obtained before and 24 hr afterwards
  Other Names: Ovidrel; r-hCG
Drug: Recombinant human follicle stimulating hormone — Recombinant human follicle stimulating hormone will be given iv and blood samples obtained before and 24 hr later.
  Other Names: Gonal-F; r-hFSH
Drug: Adrenocorticotropin — Each subject will receive a 7 hr dose-response infusion of Adrenocorticotropin.
  Other Names: Cosyntropin; ACTH
Drug: Dexamethasone — Dexamethasone will be given prior to ACTH infusion test.
  Other Names: corticosteroid
Drug: Glucose — Each subject will undergo 3 oral glcuose tolerance tests.
  Other Names: sugar

SUMMARY:
Jeffrey Chang MD is conducting a research study to learn more about the increased male hormone levels, otherwise known as androgens, seen in women with polycystic ovary syndrome (PCOS). Women with PCOS have ovaries that are comprised of many cysts, or follicles. They also have irregular or absent menstrual periods and symptoms of increased male hormones, such as facial hair or acne. In each part of the study (except part 4 which is for PCOS women only) we will be comparing responses of PCOS women to normal controls

DETAILED DESCRIPTION:
The first part of this study looks specifically at the structure of the ovaries, which are the female sex glands where both androgens and estrogens (female hormones) are made. It involves imaging your ovaries with a technology called 3-D Ultrasound. We are interested in recording the number, size and arrangement of the follicles in your ovaries.

The second part of the study looks at how the ovary produces male hormones, or androgens, with and without follicle stimulating hormone (FSH) stimulation. Hormones are substances made by a gland in one part of the body which regulate another part. FSH is a hormone naturally produced by the pituitary gland located in the brain and it helps the ovary produce estrogens, or female hormones. LH is a hormone also naturally produced by the pituitary gland and it has the ability to stimulate the ovary to make androgens. We are interested to see how much androgen your ovaries will produce in response to LH with and without FSH. To accomplish this, you will be given FSH as well as hCG, a drug that acts like LH to stimulate the ovary; FSH and hCG are approved by the Food and Drug Administration (FDA) for this investigational, off-label use.

The third part of the study looks at how much the adrenal glands contribute to the increase male hormone levels seen in PCOS. ACTH is a hormone naturally produced by the pituitary gland located in the brain and it stimulates the adrenals to make hormones. The adrenal glands are above the kidneys. They are chiefly responsible for helping the body adjust to stressful situations and work by producing cortisol and adrenaline. The adrenal glands also produce androgens, or male hormones. Previous studies have shown that some women with PCOS produce more male hormones from their adrenals. We are interested to see how much androgen your adrenal glands produce. To accomplish this, you will first be given dexamethasone, a stress steroid, to temporarily suppress your adrenal glands. You will then be given ACTH intravenously over the course of 7 hours to stimulate your adrenal glands.

The fourth part of the study is for PCOS women only and looks at how much the role of insulin contributes to the increase male hormone levels. Insulin is a hormone naturally produced by the pancreas that stimulates all of the cells in your body to take up glucose, or sugar, from the blood. Previous studies have shown that PCOS women who are more resistant to insulin, or whose cells do not take up glucose from the blood in response to insulin, make more male hormones. We are interested to see how much androgen your ovaries produce in response to LH before and after we temporarily decrease the amount of insulin in your blood. To accomplish this, you will again be given hCG, a drug that acts like LH to stimulate the ovary, with and without diazoxide, a drug that decreases the amount of insulin in your bloodstream. These tests will all be done after you are on a diet that limits how much sugar you eat. To test how much insulin you make, you will also be given Oral Glucose Tolerance Tests before and after diazoxide. This test is done by drinking a sugary liquid and testing your blood over 3 hours.

ELIGIBILITY:
Inclusion Criteria:

A group of 40 women with PCOS and 20 normal women ages 18-37 will be studied.

* Subjects will be determined to have PCOS based on clinical history of irregular menses and clinical or laboratory evidence of hyperandrogenism and polycystic ovaries on ultrasound.
* Subjects should not have been on any hormonal therapy or metformin for at least 2 months prior to study start.
* Subjects will be determined to be normal controls if they have a clinical history of regular periods

Exclusion Criteria:

* Women with hemoglobin less than 11 gm/dl at screening evaluation
* Women with untreated thyroid abnormalities
* Pregnant women or women who are nursing
* Women with BMI > 37
* Women with known sensitivity to the agents being used
* Women with prosthetic devices (i.e.,ear)/ shunts (ventricular), Hearing aids, Metal plate/pins/screws/wires
* Women with diabetes, or renal, liver, or heart disease.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2009-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Jeffrey Chang, M.D., Principal Investigator — Professor
Locations (1):
- UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from UC San Dego clinics and by advertisement in the community. Recruitment began in the summer of 2011 and was completed in Septemebr 2013. Explanation of the research protocol was done by phone and in person.
Pre-assignment Details: 41 subjects recruited. 5 dropped out prior to study. Of 36 eligible for adrenal study, 8 dropped out before study,
Groups:
- PCOS Women: Each subject will undergo pelvic ultrasound followed by iv recombinant human chorionic gonadotropin (r-hCG) stimulation. 1 month later the r-hCG test will be repeated 24 hr after injection of recombinant human follicle stimulating hormone (FSH).
  After 1 month, subjects will receive a 7 hr dose-response infusion of adrenocorticotropin (ACTH) with blood sampling. Dexamethasone will be given prior to ACTH.
  After 1 month, subject will receive r-hCG as described above followed the next day by an oral glucose tolerance test (OGTT). Subsequently, subjects will take Diazoxide 3 times a day for 2 weeks. At weekly intervals (2 weeks), the r-hCG stimulation test will be repeated followed the next day by an OGTT.
- Normal Women: Each subject will undergo pelvic ultrasound followed by iv recombinant human chorionic gonadotropin (r-hCG) stimulation. 1 month later the r-hCG test will be repeated 24 hr after an injection of recombinant human follicle stimulating hormone (FSH).
  After 1 month, subjects will receive a 7 hr dose-response infusion of adrenocorticotropin (ACTH) with blood sampling. Dexamethasone will be given prior to ACTH.
  After 1 month, subject will receive r-hCG as described above followed the next day by an oral glucose tolerance test (OGTT). Subsequently, subjects will take Diazoxide 3 times a day for 2 weeks. At weekly intervals (2 weeks), the r-hCG stimulation test will be repeated followed the next day by an OGTT.
Period: Ovarian Response to hCG
Arm/Group | PCOS Women | Normal Women
Started | 21 | 20
Completed | 18 | 18
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2
Period: Adrenal Response ot ACTH
Arm/Group | PCOS Women | Normal Women
Started | 18 (15 subjects that completed part 1 elected to participate in Part 2) | 18 (15 subjects that completed part 1 elected to participate in Part 2)
Completed | 13 (Of 18 eligible, 15 consented. 2 dropped out and 13 completed study) | 15 (Of 18 eligible, 15 consented and completed study)
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PCOS Women | Normal Women | Total
Number analyzed (Participants) | 21 | 20 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 20 | 41
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 20 | 41
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41

OUTCOME MEASURES:

1. Primary Outcome: 17-hydroxyprogesterone Responses to hCG in PCOS Women and Normal Controls
Description: Change from baseline in 17-hydroxyprogesterone at 24 hours after hCG injection
Time Frame: Baseline and 24 hours after hCG
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- NR-PCOS Women: PCOS women with normal 17-OHP responses to hCG are designated as NR-PCOS. Each subject will undergo pelvic ultrasound followed by iv recombinant human chorionic gonadotropin (r-hCG) stimulation. 1 month later the r-hCG test will be repeated 24 hr after injection of recombinant human follicle stimulating hormone (FSH).
  After 1 month, subjects will receive a 7 hr dose-response infusion of adrenocorticotropin (ACTH) with blood sampling. Dexamethasone will be given prior to ACTH.
  After 1 month, subject will receive r-hCG as described above followed the next day by an oral glucose tolerance test (OGTT). Subsequently, subjects will take Diazoxide 3 times a day for 2 weeks. At weekly intervals (2 weeks), the r-hCG stimulation test will be repeated followed the next day by an OGTT.
- HR-PCOS Women: PCOS women with exaggerated 17-OHP responses to hCG are designated as HR-PCOS. Each subject will undergo pelvic ultrasound followed by iv recombinant human chorionic gonadotropin (r-hCG) stimulation. 1 month later the r-hCG test will be repeated 24 hr after injection of recombinant human follicle stimulating hormone (FSH).
  After 1 month, subjects will receive a 7 hr dose-response infusion of adrenocorticotropin (ACTH) with blood sampling. Dexamethasone will be given prior to ACTH.
  After 1 month, subject will receive r-hCG as described above followed the next day by an oral glucose tolerance test (OGTT). Subsequently, subjects will take Diazoxide 3 times a day for 2 weeks. At weekly intervals (2 weeks), the r-hCG stimulation test will be repeated followed the next day by an OGTT.
Arm/Group | NR-PCOS Women | HR-PCOS Women | Normal Women
Number analyzed (Participants) | 10 | 8 | 18
ng/ml | 1.3 (0.2) | 3 (1) | 1.1 (0.2)

2. Secondary Outcome: Adrenal 17-hydroxyprogesterone Response to ACTH in PCOS Women and Normal Controls
Description: 17-hydroxyprogesterone response to ACTH infusion in women with PCOS and normal women. Response is reported as a single value generated by summing the data at end time frame.
Time Frame: Baseline and 1, 2, 3, 4, 5, and 6 hours after ACTH
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | NR-PCOS Women | HR-PCOS Women | Normal Women
Number analyzed (Participants) | 6 | 7 | 15
ng/ml | 6.0 (0.8) | 8.1 (0.4) | 6.2 (0.4)

3. Secondary Outcome: 17 Hydroxyprogesterone Response to hCG Injection After Lowered Insulin Levels.
Description: 17 hydroxyprogesterone levels
Time Frame: Baseline and 24 after hCG
Measure: Count of Participants; unit: Participants
Arm/Group | NR-PCOS Women | HR-PCOS Women | Normal Women
Number analyzed (Participants) | 0 | 2 | 2
Participants | 0 | 0 | 0

4. Secondary Outcome: Anti-Mullerian Hormone (AMH)
Time Frame: Baseline
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | NR-PCOS Women | HR-PCOS Women | Normal Women
Number analyzed (Participants) | 10 | 8 | 18
ng/ml | 16.0 (1.5) | 6.7 (1.5) | 5.3 (1.0)

5. Other Pre Specified Outcome: Follicle Count on 3-D Ultrasound in PCOS Women and Normal Controls
Description: 3-D ultrasound was not assessed; instead 2-D ultrasound was performed
Time Frame: baseline
Measure: Mean (Standard Error); unit: Antral Follicle Count
Arm/Group | NR-PCOS Women | HR-PCOS Women | Normal Women
Number analyzed (Participants) | 10 | 8 | 18
Antral Follicle Count | 64.4 (9.5) | 49.3 (5.6) | 31.8 (3.4)

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- PCOS Women: Each subject will undergo pelvic 3D ultrasound and an iv recombinant human chorionic gonadotropin (r-hCG) stimulation test. One month later r-hCG test will be repeated 24 hr after injection of recombinant human follicle stimulating hormone (FSH).
  After 1 month, subjects will receive a 7 hr dose-response infusion of adrenocorticotropin (ACTH) with blood sampling. Dexamethasone will be given before ACTH.
  After 1 month, subject will receive r-hCG as described above followed the next day by an oral glucose tolerance test (OGTT). Subsequently, subjects will take Diazoxide 3 times a day for 2 weeks. At weekly intervals, the r-hCG stimulation test and OGTT will be repeated as described above.
  3-D Ultrasound: One time pelvic ultrasound
  recombinant human chorionic gonadotropin: Recombinant human chorionic gonadotropin will be given iv and blood samples obtained before and 24 hr afterwards
  Recombinant human follicle stimulating
- Normal Women: Each subject will undergo pelvic 3D ultrasound and an iv recombinant human chorionic gonadotropin (r-hCG) stimulation test. One month later the r-hCG test will be repeated 24 hr after an injection of recombinant human follicle stimulating hormone (FSH).
  After 1 month, subjects will receive a 7 hr dose-response infusion of adrenocorticotropin (ACTH) with blood sampling. Dexamethasone will be given prior to ACTH.
  After 1 month, subject will receive r-hCG as described above followed the next day by an oral glucose tolerance test (OGTT). Subsequently, subjects will take Diazoxide 3 times a day for 2 weeks. At weekly intervals, the r-hCG stimulation test and OGTT will be repeated as described above.
  3-D Ultrasound: One time pelvic ultrasound
  recombinant human chorionic gonadotropin: Recombinant human chorionic gonadotropin will be given iv and blood samples obtained before and 24 hr afterwards
  Recombinant human follicle stimulati
Arm/Group | PCOS Women | Normal Women
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 0/21 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No